CLINICAL TRIAL: NCT02866448
Title: The Impact of Isoquercetin and Aspirin on Platelet Function
Brief Title: Impact of isoQUercetin and Aspirin on Platelet Function
Acronym: QUAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding delayed beyond acceptable start date
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Quercegen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Julie Lovegrove, Head of Hugh Sinclair Unit of Human Nutrition, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 16/38
Record Dates: First submitted 2016-08-02; First posted 2016-08-15 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Flavonoid; Isoquercetin; Aspirin; Platelet function; Vascular function; Blood pressure
MeSH Terms: conditions — Cardiovascular Diseases | interventions — isoquercitrin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vehicle control (Placebo Comparator): Subjects will consume
  * 4 x 250mg cellulose capsules containing 250mg cellulose, 62mg Ascorbic acid (Vitamin C), 5mg Nicotinic acid (Vitamin B3) and 0.25mg Folic Acid
  * 1 x 75mg cellulose pill
  Interventions: Drug: Vehicle control
- Isoquercetin (Experimental): Subjects will consume
  * 4 x 250mg isoquercetin capsules containing 250mg isoquercetin, 62mg Ascorbic acid (Vitamin C), 5mg Nicotinic acid (Vitamin B3) and 0.25mg Folic Acid
  * 1 x 75mg cellulose pill
  Interventions: Drug: Isoquercetin
- Aspirin (Active Comparator): Subjects will consume
  * 1 x 75mg dispersible aspirin
  * 4 x 250mg cellulose capsules containing 250mg cellulose, 62mg Ascorbic acid (Vitamin C), 5mg Nicotinic acid (Vitamin B3) and 0.25mg Folic Acid
  Interventions: Drug: Aspirin
- Isoquercetin plus Aspirin (Experimental): Subjects will consume
  * 4 x 250mg isoquercetin capsules containing 250mg isoquercetin, 62mg Ascorbic acid (Vitamin C), 5mg Nicotinic acid (Vitamin B3) and 0.25mg folic acid
  * 1 x 75mg dispersible aspirin
  Interventions: Drug: Isoquercetin plus Aspirin

INTERVENTIONS:
Drug: Vehicle control — Described in arm
  Other Names: Vehicle
  Arms: Vehicle control
Drug: Isoquercetin — Described in arm
  Other Names: IsoQ, IsoQblend
  Arms: Isoquercetin
Drug: Aspirin — Described in arm
  Other Names: ASA
  Arms: Aspirin
Drug: Isoquercetin plus Aspirin — Described in arm
  Other Names: IsoQ + ASA
  Arms: Isoquercetin plus Aspirin

SUMMARY:
The purpose of this study is to investigate the effect of acute isoquercetin supplementation, aspirin, and isoquercetin/aspirin combination on platelet aggregation, blood pressure and vasculat stiffness (eg digital volume pulse), as well as investigating the plasma accumulation and urine excretion profiles of quercetin.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide. In 2012, approximately 17.5 million people worldwide died from CVD, representing 31% of global death. Flavonoids are a class of plant secondary metabolites, functioning in the plant to aid in growth. These compounds are found in diets worldwide, and many cohort studies have demonstrated the protective effect of diets high in flavonoids against CVD events, with some studies showing flavonoid intake inversely associated with CV event risk, CV non-fatal events and all-cause mortality. One consistent issue with quercetin as a dietary flavonoid is the plasma concentrations it is able to reach are not always sufficient to provide a protective effect. Therefore, supplementation or pharmacological intervention with flavonoids may offer a solution. Supplementation with isoquercetin, the 3-O-glucoside of quercetin, offers the potential for much higher plasma concentrations of quercetin and its metabolites than dietary sources can offer, with associated increased inhibitory, anti-platelet effects. It must therefore be addressed whether isoquercetin supplementation can effectively reduce platelet function ex vivo, measured by aggregation and closure time, as well as improve vascular function, measured through blood pressure (BP) and vascular stiffness (eg digital volume pulse (DVP)).

ELIGIBILITY:
Inclusion Criteria:

* Plasma TAG (triacylglycerol) < 4.0 mmol/l
* Body mass index (BMI) between 18-35 kg/m2
* Total cholesterol (TC): <7 mmol/l
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* Consume less than 5 portions of fruit/vegetables per day
* Male

Exclusion Criteria:

* Suffered a myocardial infarction/stroke in the past 12 months
* Diabetic (diagnosed as fasting blood glucose >7 mmol/l) or suffer from other endocrine disorders
* Suffering from renal or bowel disease or have a history of cholestatic liver or pancreatitis
* On drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* History of alcohol abuse
* Planning or on a weight reducing regime
* Undertake vigorous exercise more than 3 times a week
* Taking nutritional supplements (e.g. fish oil, calcium)
* Taking flavonoid supplements
* Suffering from hayfever
* Taking any, or intolerant to, NSAIDS including aspirin
* On any medication, prescribed or not prescribed (or willing to abstain from these during period of study as well as prior 2 week washout period)
* Using any recreational drugs
* Vegan
* Intolerant/allergic to nuts, wheat, dairy
* Intolerant/allergic to aspirin
* On, or have taken antibiotics in the last 2 months
* Had surgery in the last 3 months
* Smokers, or have smoked in the last month
* Using e-cigarettes
* Anaemic: haemoglobin <12.5 g/dl
* History of gastric ulcers
* Female

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in platelet aggregation | Acute Study: measured at -60 (baseline), 120, 240 and 360min

SECONDARY OUTCOMES:
Change from baseline in Closure Time (CT), measured with a Platelet Function Analyzer (PFA) | Acute study: measured at -60 (baseline), 120, 240 and 360min
Change from baseline in blood pressure (systolic pressure, diastolic pressure and pulse pressure) | Acute study: measured at -60 (baseline), 0, 30, 60, 90, 120, 180, 240, 300 and 360min
Change from baseline in arterial stiffness measured by digital volume pulse - stiffness index | Acute study: measured at -60 (baseline), 0, 30, 60, 90, 120, 180, 240, 300 and 360min
Change from baseline in arterial stiffness measured by digital volume pulse - reflection index | Acute study: measured at -60 (baseline), 0, 30, 60, 90, 120, 180, 240, 300 and 360min
Change from baseline in total plasma quercetin concentration (micromolar) | Acute study: measured at -60 (baseline), 0, 30, 60, 90, 120, 180, 240, 300 and 360min
Change from baseline in total urine quercetin concentration (micromolar) | Acute study: measured at 0 (baseline),120, 240 and 360min

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc PhD RNutr, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be averaged (some will also be normalized) before publishing, IPD (Individual Participant Data) will not be made available